CLINICAL TRIAL: NCT06251375
Title: Sedation Practice in Intensive Care Evaluation (SPICE IV) Early Sedation With Dexmedetomidine vs. Placebo in Older Ventilated Critically Ill Patients: A Prospective, Multi-Centre, Double-Blind, Randomized, Controlled Trial
Brief Title: Early Sedation With Dexmedetomidine vs. Placebo in Older Ventilated Critically Ill Patients
Acronym: SPICEIV
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Kimberley Lewis, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4569
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Insufficiency
Keywords: Mechanical Ventilation; Sedation; Randomized Control Trial; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The SPICE IV trial is a prospective, double-blind, placebo controlled, randomised trial of early sedation with dexmedetomidine in invasively mechanically ventilated patients who are ≥ 65 years of age and who are expected to remain ventilated more than one calendar day after randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain blinding of patients, investigators, clinical staff, and research coordinators, pre-packaged study medication kits will be used. Upon randomization, the website will assign a unique study number and a unique 'medication kit number' to each participant. The unique medication kit number is matched to blinded study drug according to the patient's treatment allocation, supplied to the site. Each medication kit will contain either: dexmedetomidine 200 µg/2 ml vials or normal saline vials. Blinding of study medications within the medication kit will be achieved by identical labelled 2 ml vials.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine Intervention (Experimental): Patients randomized to the experimental arm will receive dexmedetomidine. The study medication will be reconstituted by mixing 4 vials (8 ml) into a 100 ml bag of normal saline or 5% dextrose, this is the preferred dilution, or 2 vials (4ml) into 50 ml syringe to an equivalent concentration of 8 mcg/ml of dexmedetomidine. The constituted infusion is stable at room temperature for up to 24 hours.
  The recommended starting infusion rate is equivalent to 1 µg/kg/h of dexmedetomidine, without loading or bolus. This will be titrated to an equivalent dexmedetomidine dose of 0 to 1.0 µg/kg/h according to study algorithm to maintain target sedation of Richmond Agitation-Sedation Scale (RASS) score of -1 to +1.
  Interventions: Drug: Dexmedetomidine
- Control Intervention (Placebo Comparator): Those in the control group will receive a placebo that is identical in colour and packaging and at equal volume to the intervention group. The placebo is a matching vial containing 2 mL sterile normal saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is an α2-adrenergic agonist sedative commonly used in invasive mechanical ventilation that promotes patient wakefulness, has no effect on respiratory drive, has important analgesic properties, and when compared to γ-aminobutyric acid receptor agonists like benzodiazepines, reduces delirium.
  Arms: Dexmedetomidine Intervention
Other: Placebo — Normal saline placebo will be given as continuous infusion.
  Arms: Control Intervention

SUMMARY:
Sedation remains a ubiquitous and crucial component of intensive care treatments in critically ill mechanically ventilated patients. Sedation relieves anxiety, reduces distress, and promotes tolerance of endotracheal intubation and associated life-sustaining interventions such as mechanical ventilation, cardiovascular assistance, and renal support. Thus, choosing the optimal sedative agent is vital to patient comfort, safety, and survival. Despite more than 20 years of intensive care sedation research, there is still no consensus on what constitutes best sedation practice. The Society of Critical Care Medicine, the premier critical care organisation in North America, published the 2018 Clinical Practice Guidelines on the management of Pain, Agitation/Sedation, Delirium, Immobility and Sleep (PADIS) disruption (chaired by our primary applicant W.A.) and issued weak recommendations to provide analgesia before sedation, to target light sedation whenever clinically feasible, and to use either dexmedetomidine or propofol over midazolam for the sedation of mechanically ventilated critically ill patients. Similarly, the American Thoracic Society produced a set of Clinical Practice Guidelines to promote liberation and weaning from mechanical ventilation in critically ill patients, with weak recommendations for the use of non-benzodiazepines as primary sedatives and to target light sedation when clinically possible. A weak recommendation was issued in an Intensive Care Medicine Rapid Practice Guideline published in 2022 to use dexmedetomidine over propofol for sedation of critically ill adults, if the desired outcome is a reduction in delirium. These guidelines, however, do not consider age-dependent pharmacokinetics and pharmacodynamics, illness severity, timing of sedative administration, operative vs medical reason for admission, or the changing dynamics of sedation practice at different phases of critical illness. The lack of high-level evidence to inform sedation practice in the critically ill has led to approaches that are mainly opinion-based and lack the support of evidence from large multicentre, international randomised clinical trials.

DETAILED DESCRIPTION:
1. BACKGROUND

   Current guidelines highlight evidence gaps to be addressed in future sedation trials, particularly the need for adequately powered trials to evaluate impact of sedative choice in older adults, as they have a highest overall mortality and the most common demographic to require an ICU admission of all age groups.

   Dexmedetomidine, an α2-adrenergic agonist sedative, may be the solution. The SPICE III trial, a prelude to the SPICE IV study, evaluated early sedation with dexmedetomidine versus usual care sedation in 4000 critically ill patients. The SPICE III trial identified a heterogeneity of treatment effect (HTE) on the primary outcome of 90-day mortality, suggesting lower mortality in older patients. To further evaluate the observed HTE, SPICE IV was designed as a randomized double-blind placebo-controlled trial with a study population restricted to patients at or older than 65 years of age.
2. HYPOTHESIS

   Early sedation with DEX as the primary sedative agent reduces 90-day all-cause mortality in invasively mechanically ventilated patients who are ≥ 65 years of age.
3. OBJECTIVES

   The primary aim is to determine whether, in invasively mechanically ventilated patients who are ≥ 65 years of age, early sedation with DEX as the primary sedative agent reduces 90-day all-cause mortality.

   The secondary aims are to assess the effect of DEX on ventilator free days, coma and delirium free days, major adverse kidney events (MAKE-28) at day 28, duration of ventilation, and hospital stay in survivors.
4. METHODS

This is a prospective, double-blind, placebo controlled, randomised trial of early sedation with dexmedetomidine in invasively mechanically ventilated patients who are ≥ 65 years of age and who are expected to remain ventilated more than one calendar day after randomization. Randomization will occur via a secured website. A total of 300 patients will be recruited across Canadian centres and assigned in a 1:1 ratio to either: early dexmedetomidine (Intervention arm) or placebo (Control arm).Patients in the active intervention arm will receive a dexmedetomidine infusion starting at a recommended dose of 1 µg/kg/h without a loading dose. Patients in the control arm will receive normal saline at equivalent doses. Analgesia will be optimized in both groups as clinically indicated. The sedation target is defined by the Richmond Agitation-Sedation Scale (RASS) score of -1 to +1 at all times, unless otherwise clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years
2. Intubated and receiving invasive mechanical ventilation in an intensive care unit
3. The treating clinicians believe that the patient will remain intubated and ventilated until the day after tomorrow (i.e. unlikely to be extubated the following day)
4. The patient requires immediate ongoing sedative medication for comfort, safety and to facilitate the delivery of life support measures.

Exclusion Criteria:

1. Has been intubated (excluding time spent intubated within an operating theatre or transport) for greater than 12 hours, with an additional 6-hour grace period, a total of 18 hours, in an intensive care unit
2. Proven or suspected acute primary brain lesion such as traumatic brain injury, haemorrhage, stroke, or hypoxic brain injury
3. Proven or suspected spinal cord injury or other pathology that may result in permanent or prolonged weakness
4. Admission as a consequence of a suspected or proven drug overdose or burns
5. Administration of or need for ongoing neuromuscular blockade
6. A mean arterial blood (MAP) pressure that is less than 50 mmHg, despite adequate resuscitation and vasopressor support at time of randomization
7. Heart rate less than 55 beats per minute or a high grade atrio-ventricular block in the absence of a functioning pacemaker
8. Known sensitivity to dexmedetomidine
9. Acute fulminant hepatic failure with EITHER

   1. hepatic encephalopathy OR
   2. bilirubin (>300 µmol/l) and INR (>3.5), or both, without prior hepatic dysfunction.
10. Receiving full time residential nursing care
11. Death is deemed both imminent and inevitable and either the attending physician, patient or substitute decision maker is not committed to active treatment
12. Underlying disease that makes survival to 90 days unlikely
13. Previously enrolled in the SPICE IV study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  90-day all-cause mortality

SECONDARY OUTCOMES:
Number of days alive and free of coma and delirium | 28 days
Number of days alive and ventilator free | 28 days
Major Adverse Kidney Events | 28 days
  Mortality + Acute Kidney Injury > stage II, defined by Kidney Disease Improving Global Outcome (KDIGO) definition
Duration of mechanical ventilation in survivors | 28 days
Hospital Length of Stay in survivors | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Lewis, MD, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster University
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada